CLINICAL TRIAL: NCT05400304
Title: Preoperative CT-based Radiomics Combined With Intraoperative Frozen Section is Predictive of Spread Through Air Space in Early Lung Adenocarcinoma
Brief Title: Radiomics Combined With Frozen Section Prediction Model for Spread Through Air Space in Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: RFSTAS
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Lung Adenocarcinoma
Keywords: Spread Through Air Space; radiomics; frozen section; Prediction Model
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training dataset: No interventions
  Interventions: Diagnostic Test: radiomics
- External validation1: No interventions
  Interventions: Diagnostic Test: radiomics
- External validation2: No interventions
  Interventions: Diagnostic Test: radiomics

INTERVENTIONS:
Diagnostic Test: radiomics — The high-throughput extraction of large amounts of quantitative image features from medical images

SUMMARY:
a multifactorial model combining radiomics with frozen section analysis is a potential biomarker for assessing Spread Through Air Space during surgery, which can provide decision-making support to therapeutic planning for early-stage lung adenocarcinomas.

DETAILED DESCRIPTION:
Spread through air space (STAS) is a novel invasive pattern of lung adenocarcinoma and is also a risk factor for recurrence and worse prognosis of lung adenocarcinoma. Its preoperative assessment could thus be useful to customize surgical treatment. Radiomics and frozen section haave been recently proposed to predict STAS in patients with lung adenocarcinoma. Radiomics-based Prediction Model is highly sensitive but not specific for STAS detection. While, frozen section is highly specific but not sensitive for STAS detection in early lung adenocarcinomas.

Therefore, the proposed project aims to develop and validate a multifactorial model combining radiomics with frozen section analysis to assesse Spread Through Air Space during surgery, which can provide decision-making support to therapeutic planning for early-stage lung adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

1. intraoperative frozen section diagnosis and final pathology diagnosis are available
2. preoperative standard non-enhanced CT is available
3. Pathologically confirmed

Exclusion Criteria:

1. with a previous history of radiation therapy, chemotherapy or biopsy
2. the time interval between the CT examination and surgery was more than two weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodules in the collaborating institutes.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 24 hour before operation
  Testing the sensitivity of Radiomics to predict STAS using the area under receiver operating characteristic curve
Specificity | 24 hour before operation
  Testing the specificity of Radiomics to predict STAS using the area under receiver operating characteristic curve